CLINICAL TRIAL: NCT03287804
Title: A Single-Arm, Open-Label, Multi-Centre, Phase I/II Study Evaluating the Safety and Clinical Activity of AUTO2, a CAR T Cell Treatment Targeting BCMA and TACI, in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: APRIL CAR T Cells (AUTO2) Targeting BCMA and TACI for the Treatment of Multiple Myeloma
Acronym: APRIL
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Preliminary efficacy seen to date following treatment with AUTO2 has been determined not sufficient to warrant further development
Sponsor: Autolus Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUTO2-MM1; 2016-003893-42 (EudraCT Number)
Record Dates: First submitted 2017-09-11; First posted 2017-09-19 (Actual); Results first posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-09

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Relapsed Multiple Myeloma; Refractory Multiple Myeloma; AUTO2
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AUTO2 (Experimental): Relapsed or refractory Myeloma patients
  Interventions: Biological: AUTO2

INTERVENTIONS:
Biological: AUTO2 — AUTO2 (APRIL CAR T Cells) Following preconditioning with chemotherapy (cyclophosphamide and fludarabine) patients will be treated with doses from 15 x 10⁶ to 350 x 10⁶ APRIL CAR T Cells.
  Following Phase 2 dose determination patients will be treated with selected dose of APRIL CAR T Cells

SUMMARY:
The purpose of this study is to test the safety and efficacy of AUTO2, a CAR T Cell Treatment Targeting BCMA and TACI, in Patients with Relapsed or Refractory Multiple Myeloma.

DETAILED DESCRIPTION:
The study will consist of 2 phases, a Phase I/dose escalation phase and a Phase II/expansion phase. Patients with relapsed and relapsed or refractory multiple myeloma will be enrolled in both phases of the study. Eligible patients will undergo leukapheresis in order to harvest T cells, which is the starting material for the manufacture of the autologous CAR T product AUTO2. AUTO2 has a dual target BCMA (B cell maturation antigen) and TACI (Transmembrane activator and calcium modulator and cyclophilin ligand interactor). Following pre-conditioning by a chemotherapeutic regimen, the patient will receive AUTO2 intravenously as a single or split dose and will then enter a 12-month follow-up period.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female patients, aged ≥ 18.
2. Willing and able to give written, informed consent.
3. Confirmed diagnosis of MM.
4. Measurable disease as defined by IMWG.
5. Relapse or refractory disease and have had at least 3 different prior lines of therapy including proteasome inhibitor, alkylator and immunomodulatory therapy (IMiD), or have "double refractory" disease to a proteasome inhibitor and IMiD.
6. For females of childbearing potential, a negative serum or urine pregnancy test must be documented at screening and confirmed before receiving study treatment.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 1.
8. Peripheral blood total lymphocyte count > 0.5 x 10⁹/L.

Key Exclusion Criteria:

1. Women who are pregnant or lactating.
2. Prior treatment with investigational or approved gene therapy or cell therapy products.
3. Patient has previously received an allogenic stem cell transplant.
4. Clinically significant, uncontrolled heart disease or a recent (within 6 months) cardiac event.
5. Left Ventricular Ejection fraction < 50 unless the institutional lower limit of normal is lower.
6. Significant liver disease: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 3 × ULN, or total bilirubin > 2.0 mg/dL or evidence of end stage liver disease (e.g. ascites, hepatic encephalopathy).
7. Chronic renal impairment requiring dialysis, or calculated creatinine clearance < 30 mL/min
8. Active infectious bacterial or viral disease (hepatitis B virus, hepatitis C virus, human immunodeficiency virus, human T-lymphotropic virus or syphilis) requiring treatmenUse of rituximab within the last 3 months.
9. Active autoimmune disease requiring immunosuppression.
10. Received any anti-myeloma therapy within the last 21 days prior to preconditioning or 10 days prior to leukapheresis; steroids of up to 160 mg of dexamethasone are permitted so long as > 7 days post-dose prior to pre-conditioning or leukapheresis.
11. Known allergy to albumin, dimethyl sulfoxide (DMSO), cyclophosphamide or fludarabine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Autolus Limited, Study Director — Sponsor GmbH
Locations (4):
- VU University Medical Centre Amsterdam, Amsterdam, Netherlands
- United Kingdom (3):
  - University College London Hospitals NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Freeman Hospital, The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne

REFERENCES:
- [Derived] Lee L, Lim WC, Galas-Filipowicz D, Fung K, Taylor J, Patel D, Akbar Z, Alvarez Mediavilla E, Wawrzyniecka P, Shome D, Reijmers RM, Gregg T, Wood L, Day W, Cerec V, Ferrari M, Thomas S, Cordoba S, Onuoha S, Khokhar N, Peddareddigari V, Al-Hajj M, Cavet J, Zweegman S, Rodriguez-Justo M, Youg K, Pule M, Popat R. Limited efficacy of APRIL CAR in patients with multiple myeloma indicate challenges in the use of natural ligands for CAR T-cell therapy. J Immunother Cancer. 2023 Jun;11(6):e006699. doi: 10.1136/jitc-2023-006699. PMID 37399355

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Following preconditioning with chemotherapy (cyclophosphamide and fludarabine) patients were treated with doses from 15 x 10⁶ to 350 x 10⁶ APRIL CAR T Cells.
Pre-assignment Details: Screening procedures were performed up to 12 weeks before study treatment administered
Period: Overall Study
Arm/Group | AUTO2
Started | 12
Leukaperesed | 12
Started Pre-conditioning Therapy | 11
Received Study Treatment | 11
Completed | 1
Not Completed | 11
Not completed — Death | 1
Not completed — Physician Decision | 2
Not completed — Progressive disease | 8

BASELINE CHARACTERISTICS:
Arm/Group | AUTO2
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 1
  United Kingdom | 11

OUTCOME MEASURES:

1. Primary Outcome: Phase I - Number of Subjects With Grade 3 to 5 Toxicity During the Dose Limiting Toxicity (DLT) Period
Time Frame: Up to 28 days post-infusion
Population: Patients who received at least 1 dose (complete or partial) of AUTO2 therapy (infused set)
Measure: Count of Participants; unit: Participants
Arm/Group | AUTO2
Number analyzed (Participants) | 11
Participants | 0

2. Primary Outcome: Phase I - Number of Subjects With a Dose Limiting Toxicity (DLT)
Description: Dose limiting toxicity was defined as:
  Any new non-hematological AE of Grade 3 or higher toxicity using the NCI CTCAE (Version 4.03), which is probably or definitely related to AUTO2 therapy, which occurs within the DLT evaluation period, and which fails to resolve to Grade 2 or better within 14 days, despite appropriate supportive measures; A Grade 4 CRS; Any other reason for activation of the safety switch after receiving AUTO2; Any other fatal event (Grade 5) or life-threatening event (Grade 4) that cannot be managed with conventional supportive measures or which in the opinion of the SEC necessitates dose reduction or other modification to trial treatment to avoid a similar hazard in future patients. Effort should be made to perform an autopsy in case of fatal event where the aetiology is unclear; Any event that in the opinion of treating investigators and/or Medical Monitor puts the patient at undue risk may also be considered a DLT.
Time Frame: Up to 28 days post-infusion
Measure: Count of Participants; unit: Participants
Arm/Group | AUTO2
Number analyzed (Participants) | 11
Participants | 0

3. Primary Outcome: Number of Infused Patients With Best Overall Response
Description: Best overall response was defined as stringent complete response + complete response + very good partial response + partial response following treatment with AUTO2. Response Criteria Per IMWG Consensus Recommendations
Time Frame: Up to 2 years
Population: All patients who received at least 1 dose (complete or partial) of AUTO2 therapy in Phase I of the study were included in this analysis. No patients were enrolled in Phase II as the study was early terminated in Phase I. 2 patients were retreated; their best overall response is presented for this endpoint
Measure: Count of Participants; unit: Participants
Arm/Group | AUTO2
Number analyzed (Participants) | 11
Participants | 4

4. Secondary Outcome: Proportion of Patients for Whom an AUTO2 Product Can be Generated
Description: Feasibility of product generation was examined by assessing the number of AUTO2 successfully manufactured as a fraction of the number of patients undergoing leukapheresis (all patients registered).
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | AUTO2
Number analyzed (Participants) | 12
Participants | 12

5. Secondary Outcome: Clinical Benefit Rate
Description: Number of subjects exhibiting stringent complete response, complete response, very good partial response, partial response or minor response following treatment with AUTO2
Time Frame: Up to 2 years
Population: All patients who received at least 1 dose (complete or partial) of AUTO2 therapy in Phase I of the study were included in this analysis. 2 patients were retreated; their best overall response is presented for this endpoint
Measure: Count of Participants; unit: Participants
Arm/Group | AUTO2
Number analyzed (Participants) | 11
Participants | 4

6. Secondary Outcome: Duration of Response
Description: Calculated from the date of first observation of sCR, CR, VGPR or PR to the date of disease progression, relapse or death, for patients who were considered responders (achieved at least PR). Patients who had not progressed, relapsed or died will be censored at the last adequate disease assessment.
Time Frame: Up to 2 years
Population: Analysis was not performed due to not enough patients who had a response (VGPR, PR) to justify the duration of response. The study was terminated early and Phase 2 was not started.
Arm/Group | AUTO2
Number analyzed (Participants) | 0

7. Secondary Outcome: Time to Disease Progression
Description: Calculated from the date of AUTO2 treatment to the date of progression. Patients who had not progressed, relapsed or died without progression/relapse will be censored at the last adequate disease assessment.
Time Frame: Up to 2 years
Population: Analysis was not performed due to not enough patients who had a response (VGPR, PR) to justify the time to disease progression. The study was terminated early and Phase 2 was not started.
Arm/Group | AUTO2
Number analyzed (Participants) | 0

8. Secondary Outcome: Progression-free Survival
Description: Calculated from the date of AUTO2 treatment to the date of progression or death. Patients who have not progressed or relapsed was censored at the last adequate disease assessment
Time Frame: Up to 2 years
Population: Analysis was not performed due to not enough patients who had a response (VGPR, PR) to justify the progression-free survival. The study was terminated early and Phase 2 was not started.
Arm/Group | AUTO2
Number analyzed (Participants) | 0

9. Secondary Outcome: Overall Survival
Description: Descriptive analysis based on number of patients alive at database lock (1-May-2020).
Time Frame: Up to 2 years
Population: All patients who receive at least 1 dose (complete or partial dose) of AUTO2 therapy
Measure: Count of Participants; unit: Participants
Arm/Group | AUTO2
Number analyzed (Participants) | 11
Participants | 3

10. Secondary Outcome: Number of Patients With Expansion Followed by Persistence of RQR8/APRIL CAR Positive T Cells in the Peripheral Blood
Description: Expansion and persistence of RQR8/APRIL CAR positive T cells as determined by quantitative polymerase chain reaction and/or flow cytometry.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | AUTO2
Number analyzed (Participants) | 11
Participants | 9

ADVERSE EVENTS:
Time Frame: From Day 0 until Day 60 post last AUTO2 infusion.
Arm/Group | AUTO2
All-Cause Mortality (participants affected / at risk) | 8/11
Serious Adverse Events (participants affected / at risk) | 6/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AUTO2 (N=11)
Neutrophil count decreased (Investigations) | 1 (1)
Metaplastic breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hedache (Nervous system disorders) | 1 (1)
Pyrexia (General disorders) | 2 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AUTO2 (N=11)
Haematoma (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 (1)
Catheter site bruise (General disorders) | 1 (1)
Chills (General disorders) | 4 (4)
Fatigue (General disorders) | 6 (10)
Oedema peripheral (General disorders) | 3 (4)
Pyrexia (General disorders) | 6 (8)
Hallucination (Psychiatric disorders) | 1 (1)
ALT increased (Investigations) | 1 (1)
AST increased (Investigations) | 1 (1)
Blood ALP increased (Investigations) | 1 (1)
Blood creatinine phosphokinase increased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (2)
Neutrophil count decreased (Investigations) | 7 (71)
Platelet count decreased (Investigations) | 2 (12)
Respiratory syncytial virus test positive (Investigations) | 1 (1)
Serum ferritin increased (Investigations) | 1 (3)
Anaemia (Blood and lymphatic system disorders) | 9 (31)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (29)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (6)
Paraesthesia (Nervous system disorders) | 2 (2)
Tension headache (Nervous system disorders) | 1 (1)
Ear disorder (Ear and labyrinth disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 5 (6)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3)
Stomatitis (Gastrointestinal disorders) | 3 (3)
Micturition urgency (Renal and urinary disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (6)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (2)
Enterovirus infection (Infections and infestations) | 1 (1)
External ear cellulitis (Infections and infestations) | 1 (1)
Metapneumovirus infection (Infections and infestations) | 1 (2)
Parvovirus B19 infection (Infections and infestations) | 1 (1)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of patients analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/04/NCT03287804/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/04/NCT03287804/SAP_001.pdf